CLINICAL TRIAL: NCT02481999
Title: Pre- and Postoperative EEG-Monitoring for Children Aged From 0,5 to 8 Years
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: Narco-Kids
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia
Keywords: Depth of anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Patients: 470 children for elective surgery 0,5 to 8 years
  Analysis of EEG data will divided in four age-related groups because of the different baseline EEG activity:
  * 0.5 - 12 month: 5-7 Hz activity / blocked by eye opening
  * 12 - 36 month: 7-8 Hz activity / Variability 5 - 10 Hz
  * 3 - 6 years: 8 Hz activity / amplitude 100µV
  * 6 - 8 years 10Hz activity / amplitude 100 µV
- Control group: Healthy children for POCD assessment: 80 healthy children (siblings of study group children and children from Kindergarten) 0,5 to 8 years with no operation

SUMMARY:
Evaluation of mechanisms and factors of anaesthesia on postoperative delirium and emergence agitation as well as on postoperative cognitive function in children aged 0,5-8 years scheduled for elective surgery. The depth of anesthesia in children for elective surgery aged 0,5-6 years is monitored with intraoperative "Narcotrend-Compact-M-Monitoring". Postoperatively the "Pediatric Anesthesia Emergence Delirium Scores (PAED Score)" [Sikich et al. 2004;Locatelli et al. 2013] is used to screen for the frequency of postoperative delirium in the post anesthesia care unit discharge of the child after surgery. Cognitive testings are performed in children of the study group (n= 470) and a control group (n= 80) with the parents support to evaluate deficits in children in their cognitive areas (POCD (Postoperative cognitive deficit)) at three different time points up to three months.

DETAILED DESCRIPTION:
According to recent studies in children aged from 0,5 to 8 years "Narcotrend Monitor" (from EEG derived monitoring of the frontal brain waves) can reliably measure the depth of anesthesia [Münte et al. 2009; Weber et al. 2005].

Depth of anesthesia in adults is significantly correlated with the incidence of postoperative delirium and longer lasting cognitive deficits [Radtke et al. 2013; Chan et al. 2013; Whitlock et al. 2014].

We know from animal experimental studies that anesthetics have a potential toxic effect in the developing brain. [Sinner et al 2014].

After two years (approximately 1/3 - 1/2 of the total sample) an interim analysis with recalculation of the case numbers is carried out, if the initial effect sizes differ strongly.

ELIGIBILITY:
Study Group.

Inclusion Criteria:

* male or female children 0,5 to 8 years
* planned elective surgery
* informed consent by both parents, if both parents have joint custody

Exclusion Criteria:

* indication for isolation of patients with multi-resistant bacteria
* known neurological or psychiatric precondition (disease)
* inability of the parents to speak and or read German
* lacking willingness to save and hand out pseudonomized data within the clinical study
* contact allergy to silver or silver chloride
* participation in another prospective interventional clinical study during this study

Control Group:

Inclusion Criteria:

* male or female healthy children 0,5 to 8 years (siblings of study group and children from kindergarten)
* no planned operation in the next three month
* no operation in the last half year before study inclusion
* informed consent by both parents, if both parents have joint custody

Exclusion Criteria:

* Neurological or psychiatric precondition (disease), which limits the conduction of the neurocognitive testing
* Anacusis or Hypoacusis, which limits the conduction of the neurocognitive testing
* Taking psychotropic drugs (including sleep-inducing drug and benzodiazepine) on a regular basis and substances, which limit the conduction of the neurocognitive testing
* Inability of the parents to speak and or read the used language
* Lacking willingness to save and hand out pseudonomized data within the clinical study

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children for elective surgery aged from 0, 5 to 8 years
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence delirium and postoperative delirium | Until discharge of the child from the recovery room, an expected average of 1 hour
  The Delirium is measured by the Pediatric Anesthesia Emergence Delirium Scores (PAED Score) (Sikich et al. 2004; Locatelli et al. 2013)

SECONDARY OUTCOMES:
Depth of anesthesia | During the operation
  Depth of anesthesia assessed by band-power of the 4 frequency bands (alpha, beta, theta, delta) and activity in percentages of total spectral power ( F50% / F95%) assessed with Narcotrend Monitor
Incidence of behavioral problem | Up to 5 postoperative days
  The behavioral problem is measured by a modified Version of the Posthospital Behavior Questionnaire" (PHBQ) (Buehrer et al. 2014)
Severity of emergence Delirium | Until discharge of the child from the recovery room, an expected average of 1 hour
  The Delirium is measured by Pediatric Anesthesia Emergence Delirium Scores (PAED Score) (Sikich et al. 2004; Locatelli et al. 2013)
Duration of emergence Delirium | Until discharge of the child from the recovery room, an expected average of 1 hour
  The Delirium is measured by Pediatric Anesthesia Emergence Delirium Scores (PAED Score)" [Sikich et al. 2004; Locatelli et al. 2013]
Lactate | Up to 5 postoperative days
  Laboratory parameter
Hemoglobin | Up to 5 postoperative days
  Laboratory parameter
Soluble Interleukin - 6 | Up to the end of the operation
  Laboratory parameter
Analgesia | Up to the end of stay in the recovery room, an expected average of 1 hour
Hypnotics | Begin of Anesthesia up to the end of stay in the recovery room, an expected average of 1 hour
Stress reducing agents | Up to the end of stay in the recovery room, an expected average of 1 hour
Psychoactive drugs/Benzodiazepines | From 1h before surgery start up to the end of stay in the operation (an expected average of 2 hours)
Fluid and transfusion therapy | From one day before surgery start up to the end of stay in the recovery room (an expected average of 2 hours
  The fluid and transfusion therapy is measured by preoperative sobriety times by intraoperative fluid and volume administration and balance.
Postoperative cognitive deficit (POCD) in children 6 to 42 months | Up to 365 postoperative days
  POCD is measured by parent questionnaires (BRIEF-P) and in children by the Bayley III Scales of Infant and Toddler Development (cognitive, language, motor function and processing speed, social emotional scale) and NEPSY II (Statue, word generation, Visuomotor precision from 3 years).
Postoperative cognitive deficit (POCD) in children 43 to 96 months | Up to 365 postoperative days
  POCD is measured by parent questionnaires (BRIEF-P, BRIEF) and in children by the Colored Progressive Matrices (CPM), the CANTAB test battery and NEPSY-II subtests (Visuomotor precision, word generation, statue (until 6 years); animal sorting (from 7 years)).
Duration of anesthesia | During the operation
  Measured by Narcotrend monitor
Burst suppression ratio | During the operation
  Measured by Narcotrend monitor
Duration of surgery | During the operation
Time schedule for intraoperative EEG recording | During the operation
  Predefined time points: Baseline, start of anesthetic administration (STARTAnesth), start of analgesic administration (STARTAnalg), Loss of consciousness (LOC), airway device insertion [INT], skin incision/ surgery start (SKIN), intraoperative steady state (OP), stop of anesthetic administration (ENDAnesth), stop of analgesic administration (ENDAnalg),airway device removal [EXE] regain of consciousness (ROC), awakening (AWK)
Pain in children < 4 years | Up to the end of stay in the recovery room, an expected average of 1 hour
  Pain is measured by the FLACC- Scale
Pain in children < 4 years | Up to the end of stay in the recovery room, an expected average of 1 hour
  Pain is measured by the KUSS-Score
Pain in children ≥ 4 years | Up to the end of stay in the recovery room, an expected average of 1 hour
  Pain is measured by the Faces Pain Scale - revised
C-reactive protein | Up to 5 postoperative days
Carbon dioxide (CO2) and oxygen (O2) monitoring | During the operation
Positive endexpiratory pressure | During the operation
Inspiratory pressure | During the operation
Tidal volume breathing frequency | During the operation
Minute volume | During the operation
Anxiety of the children | Up to 365 postoperative days
  Observation of anxiety during psychological assessment on a 4-point-Likert-scale
Anxiety of the parents | Up to 365 postoperative days
  Baseline (STAI) after 3 months (STAI)
Compliance of the children | At the beginning of the operation
  Measured by Induction compliance checklist
Stress | Up to 365 postoperative days
  Stress is measured of of parents and of children. Parenting stress index (PSI) (German version: Eltern-Belastungsinventar (EBI))
Glucose | Up to 5 postoperative days
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 1 day
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Postoperative organ complications | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Behavioral changes of the children | Up to 5 postoperative days
  Post Hospitalization Behavior Questionnaire (PHBQ)
Anxiety of children | At the beginning of the operation
  mYale-SF (2-8 years)
Blood pressure | During the operation
  This Monitoring of the blood pressure will be measured at the defined EEG measurement timepoints from STARTAnesth to EXE.
Body temperature | During the operation
  This Monitoring of body temperature will be measured at the defined EEG measurement timepoints from STARTAnesth to EXE.
Heart rate | During the operation
  This Monitoring of heart rate will be measured at the defined EEG measurement timepoints from STARTAnesth to EXE.
Clinical routine anesthesia parameters | Up to the end of stay in the recovery room, an expected average of 1 hour
  Clinical routine anesthesia parameters are measured by primary induction technique, type of induction, type of maintenance of anesthesia, airway management, additional regional anesthesia, type of regional anesthesia, time of regional anesthesia, application during operation and blood gas analysis) during anesthesia until end of recovery room stay.
Blood gas analysis | Up to the end of stay in the recovery room, an expected average of 1 hour
Incidence of Delirium | Up to the end of stay in the recovery room, an expected average of 1 hour
  Incidence of Delirium is measured with the CAPD-Score [Dill et al. 2016]
Type of surgery | During the operation
Specific field of surgery | During the operation

OTHER OUTCOMES:
Age | At the beginning of the investigation
  Age will be measured in months and in years
ASA classification | At the beginning of the investigation
Medical history | At the beginning of the investigation
Previous number of surgeries | At the beginning of the investigation
Previous medication | At the beginning of the investigation
Main diagnosis | At the beginning of the investigation
  he diagnosis that is responsible for occasioning the performance of inpatient treatment.
Demographic and background data | At the beginning of the investigation
  Demographic and background data are collected by gender, ethnicity, education of the parents, language, number of siblings, family Situation)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - University Medicine Berlin, Berlin, Germany

REFERENCES:
- [Derived] Koch S, Stegherr AM, Rupp L, Kruppa J, Prager C, Kramer S, Fahlenkamp A, Spies C. Emergence delirium in children is not related to intraoperative burst suppression - prospective, observational electrography study. BMC Anesthesiol. 2019 Aug 8;19(1):146. doi: 10.1186/s12871-019-0819-2. PMID 31395011
- [Derived] Koch S, Rupp L, Prager C, Wernecke KD, Kramer S, Fahlenkamp A, Spies CD. Emergence delirium in children is related to epileptiform discharges during anaesthesia induction: An observational study. Eur J Anaesthesiol. 2018 Dec;35(12):929-936. doi: 10.1097/EJA.0000000000000867. PMID 30113351
- [Derived] Koch S, Rupp L, Prager C, Morgeli R, Kramer S, Wernecke KD, Fahlenkamp A, Spies C. Incidence of epileptiform discharges in children during induction of anaesthesia using Propofol versus Sevoflurane. Clin Neurophysiol. 2018 Aug;129(8):1642-1648. doi: 10.1016/j.clinph.2018.05.013. Epub 2018 Jun 8. PMID 29913339